CLINICAL TRIAL: NCT02602392
Title: Online Asthma Self-Management for Children Aged 5-10 and Their Parents
Acronym: ChildAsthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oregon Center for Applied Science, Inc. (Industry)
Responsible Party: Principal Investigator, Susan Schroeder, Research Scientist, Oregon Center for Applied Science, Inc.
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: SBIR77R-2RR; R44HL077965-02A2 (NIH)
Record Dates: First submitted 2013-05-31; First posted 2015-11-11 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2015-11

CONDITIONS: Asthma
Keywords: Self management; Education; Children; Caregivers; Health Care Providers
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lungtropolis (Experimental): A game-based website for children with asthma aged 5-10 to teach basic self-management skills and a comprehensive adjunct informational website for parents
  Interventions: Behavioral: Lungtropolis
- Asthma educational booklet (Active Comparator): Text-based asthma education booklet for parents and children in PDF format
  Interventions: Behavioral: Asthma educational booklet

INTERVENTIONS:
Behavioral: Lungtropolis — A game-based website for children with asthma aged 5-10 to teach basic self-management skills and a comprehensive adjunct informational website for parents
  Arms: Lungtropolis
Behavioral: Asthma educational booklet — Text-based asthma education booklet for parents and children in PDF format
  Arms: Asthma educational booklet

SUMMARY:
The potential benefits of this research to public health include improved understanding of cultural factors in pediatric asthma self-management, improved self-management skills for children, and better asthma management skills for their parents. This could result in eased suffering and improved quality of life for millions of children and their families, and also reduce the economic burden borne by society in the forms of medical expenditures and lost productivity.

DETAILED DESCRIPTION:
This proposal will create an interactive multimedia (IMM) program designed to support the self-management efforts of asthmatic children aged 5-10 years and their families. This behavior change program will be designed to promote self-management by (a) increasing child and caregiver knowledge about asthma, (b) encouraging compliance with medication protocols and environmental controls, and (c) increasing self-efficacy to create and implement an Asthma Action Plan.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 5-10 with physican-diagnosed asthma and who had been prescribed any type of asthma medication, and one of their parents or primary caregivers. Parents and children needed to have access to an internet- and video-capable computer, and the parent needed to have a valid e-mail address in order to receive study-related correspondence.

Exclusion Criteria:

* Only English-speaking participants were accepted because the program was developed only for English speakers. Children less than 5 years of age and older than 10 were excluded because the program is developed targeted to the developmental abilities and interests of children aged 5-10. There were no exclusions based on race/ethnicity.

Ages: 5 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 622 (Actual)
Dates: Start 2011-01; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in children's knowledge about asthma | 45 days
  A 5-item knowledge scale was developed with program-specific questions regarding asthma physiology, response to worsening symptoms, and asthma medications. These items used a 3-response choice scheme: "true," "not true," and "I don't know." The total number of items correct was summed to form the knowledge scale.
Change from baseline in parents' knowledge about asthma | 45 days
  The Parent Knowledge Questionnaire (alpha = .81; Mesters, et al., 2003) was adapted to match program content, creating a 19-item knowledge scale covering basic knowledge about asthma (e.g., response to worsening symptoms, asthma medications, asthma triggers). The total number of correct items was summed to form the knowledge scale.
Change from baseline in children's attitudes toward medication | 45 days
  A 5-item knowledge scale was developed with program-specific questions regarding asthma physiology, response to worsening symptoms, and asthma medications. These items used a 3-response choice scheme: "true," "not true," and "I don't know." The total number of items correct was summed to form the knowledge scale.
Change from baseline in parents' attitudes about asthma self-management | 45 days
  The Asthma Attitude Survey (Mesters, et al., 2003), adapted to fit program content, assessed parents' attitudes regarding recognition of worsening symptoms, asthma medications, and triggers management. A 5-point Likert-type scale ranging from 1 (strongly agree) to 5 (strongly disagree) was used for responses, and items were summed to create an overall attitudes score.
Change from baseline in children's self-efficacy to improve asthma self-management | 45 days
  Three self-efficacy items addressed each child's confidence in being able to recognize warning signs, use his/her quick-relief medicine immediately when having warning signs, and take medications as directed. Response choices were presented on a Likert-type scale ranging from 1 (no way, I can't do that) to 4 (sure, I can do that).
Change from baseline in parents' self-efficacy to improve asthma self-management | 45 days
  The Parent Asthma Self-Efficacy survey (Bursch, et al., 2003), adapted to fit program content, used a 5-point Likert-type scale ranging from 1 (not at all sure) to 5 (completely sure) to assess parents' confidence about administering medications and responding to worsening symptoms.

SECONDARY OUTCOMES:
Change from baseline in Asthma Control Test | 45 days
  The Child-Asthma Control Test (C-ACT) for children 4-11 years old (Nathan, et al., 2004) was used to assess the child's current level of asthma control. The C-ACT contains 7 items-4 for the child's response and 3 for the parent's response, summed to create an asthma control score. Response choices for the children were presented on a 4-point Likert-type scale. The 3 parent items asked for frequency of symptoms over the past 4 weeks and were presented on a 6-point scale.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Schroeder, MPH, MCHES, Principal Investigator — Oregon Center for Applied Science
Locations (1):
- Oregon Center for Applied Science, Eugene, Oregon, United States

REFERENCES:
- See also: Portal page from which to access the child's asthma game and the parent's informational website — http://lungtropolis.com